CLINICAL TRIAL: NCT07032103
Title: A Prospective Study for Patients With Lymphoma at the Samsung Medical Center
Brief Title: Prospective Cohort Study for Lymphoma: Samsung Lymphoma Cohort Study IV
Acronym: SMCLYM-IV
Status: Recruiting | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Kim, Seok Jin, Professor, Samsung Medical Center
Other Study IDs: SMC-Lym-IV
Record Dates: First submitted 2025-06-13; First posted 2025-06-22 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Lymphoma
Keywords: lymphoma; prognosis
MeSH Terms: conditions — Lymphoma | interventions — Palliative Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — Serum and cell-free DNA from patients' peripheral blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Immunochemotherapy — Systemic chemotherapy with curative intent
  Other Names: Supportive treatment

SUMMARY:
This prospective study enrolls patients who are diagnosed with aggressive lymphoma including Hodgkin and non-Hodgkin lymphomas. Enrolled patients will be treated according to our institution' treatment policy in clinical practice. The disease status including response to therapy and survival status will be regularly updated during the study period. Patients' serum and cell-free DNA will be collected and analyzed.

DETAILED DESCRIPTION:
The study population is aggressive lymphomas requiring systemic chemotherapy. Newly diagnosed or relapsed/refractory patients can be enrolled into the study. Patients can be treated according to the principle of routine care of our institute. The study process is as follows.

1. Registration after informed consent.
2. Laboratory and radiological evaluation after registration including collection of serum and cell-free DNA from patients' peripheral blood
3. Interim and final response evaluation including collection of serum and cell-free DNA from patients' peripheral blood
4. Regular monitoring disease status and update of survival status
5. Laboratory and radiological evaluation after relapse or progression including collection of serum and cell-free DNA from patients' peripheral blood

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically diagnosed Hodgkin and non-Hodgkin lymphomas
2. 20 years
3. Patients requiring systemic chemotherapy with curative intent
4. Written informed consent

Exclusion Criteria:

1. Myeloid malignancy
2. Multiple myeloma
3. Patients do not require systemic chemotherapy with curative intent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients are diagnosed with aggressive lymphoma including Hodgkin and non-Hodgkin lymphoma. All patients should receive systemic chemotherapy. Newly diagnosed or relapsed/refractory patients can be enrolled
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2028-12-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Reponse rate | 3 months after the completion of treatment
  Repsonse to the ist line treatment
Response | 3 months after chemotherapy
  response to treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No